CLINICAL TRIAL: NCT04885855
Title: Efficacy and Safety of 8- Versus 12-week Sofosbuvir-ravidasvir Treatment of Non-cirrhotic Chronic Hepatitis C Patients: An Open-label, Randomized, Multicenter Study in Malaysia
Brief Title: 8- Versus 12-week of Sofosbuvir-ravidasvir Treatment of Chronic Hepatitis C
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Muhammad Radzi Abu Hassan (Other Government)
Responsible Party: Sponsor-Investigator, Muhammad Radzi Abu Hassan, Consultant Gastroenterologist, Hospital Sultanah Bahiyah
Organization: Hospital Sultanah Bahiyah (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOH-8v12-SOF/RDV-01-HCV
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; ravidasvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8-week (Experimental): Patient will be receiving treatment of tablet Sofosbuvir 400mg and tablet Ravidasvir 200mg combination once daily for the duration of 8 weeks.
  Interventions: Drug: Sofosbuvir 400 MG; Drug: Ravidasvir 200mg
- 12-week (Active Comparator): Patient will be receiving treatment of tablet Sofosbuvir 400mg and tablet Ravidasvir 200mg combination once daily for the duration of 12 weeks.
  Interventions: Drug: Sofosbuvir 400 MG; Drug: Ravidasvir 200mg

INTERVENTIONS:
Drug: Sofosbuvir 400 MG — Sofosbuvir is a direct-acting antiviral (DAA) a nucleotide analog inhibitor of hepatitis C virus nonstructural protein 5B (NS5B)
  Other Names: Grateziano
Drug: Ravidasvir 200mg — Ravidasvir is an investigational direct-acting antiviral (DAA) a nucleotide analog inhibitor of hepatitis C virus nonstructural protein 5A (NS5A)
  Other Names: PPI-668

SUMMARY:
This is open-label, randomized, multicentre study to compare the efficacy and safety of the 8-week versus 12-week of SOF-RVD combination treatment for non-cirrhotic chronic hepatitis C patients.

All the recruited subjects will receive the treatment accordingly and be followed up for 24 weeks following the completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Has evidence of chronic HCV infection, defined as:

   a. Positive anti-HCV antibody or detectable HCV RNA or HCV genotype and HCV viral load ≥104 IU/mL within 6 months prior to the time of blood collection for screening.
2. Willing and able to provide written informed consent.
3. Men and women age ≥ 18 years and < 70 years.
4. Body Mass Index (BMI) of 18 to 35 kg/m2.
5. Intention to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.
6. Women with a negative pregnancy test at screening and baseline assessment.
7. Women of childbearing potential who accept effective contraception from 2 weeks prior to day 1 of study to 1 month after treatment (double contraceptive method including at least one barrier method). A woman is of non-childbearing potential if she (a) reached natural menopause determined retrospectively after 12 months of amenorrhea without any other obvious medical cause or (b) had procedures like bilateral tubal ligation or hysterectomy or bilateral oophorectomy.
8. Subjects who are compliant in opioid substitution maintenance program may be included as long as there is no concern about study medications adherence and interaction or compliance to study schedules.
9. HIV/HCV co-infected patients receiving cART fulfilling the below criteria are eligible for the study:

   1. Antiretroviral therapy has been initiated at least 6 months prior to screening (to avoid the possibility of Immune reconstitution inflammatory syndrome - IRIS)
   2. Patient has been on the same protocol-approved ARV regimen for ≥ 8 weeks prior to screening and is expected to continue the current ARV regimen through the end of study.
   3. HIV ARVs: agents allowed in this study should be administered per the prescribing information in the package insert
   4. Screening HIV RNA <50 copies/mL.
   5. Screening CD4 cell count ≥100 cells/uL
10. HIV/HCV co-infected patients not receiving cART: Screening CD4 cell count must be ≥ 500 cells/uL

Exclusion Criteria:

1. Has evidence of liver cirrhosis in which, liver cirrhosis is determined by;

   1. APRI score of ≥ 1.5,
   2. In case where APRI score is >1.0 but <1.5,

      * Perform fibroscan* (where TE ≥12.5 kPa indicates liver cirrhosis) or
      * Calculate FIB-4 index (where ≥3.25 indicates liver cirrhosis) *Depending on availability at facility
   3. Current/past history of decompensation including ascites, variceal bleeding, bacterial peritonitis, or hepatic encephalopathy.
2. Additional laboratory exclusion criteria:

   1. Direct bilirubin >3x ULN
   2. AST, ALT >10x ULN
   3. Low neutrophil count (≤599 cells/mm3), haemoglobin (<9.0 g/dL), platelets (<150000 cells/mm3).
3. Patients with serum creatinine >1.5 ULN or end-stage renal disease.2
4. Hepatitis B co-infection (HBsAg positive).
5. Pregnancy, as documented by positive pregnancy tests at screening and baseline assessment.
6. Breastfeeding.
7. Subjects currently receiving or unable to stop the use for at least 1 week prior to receiving the first dose of study drug any medications or herbal supplements known to be potent inhibitors or moderate inducers of cytochrome P450 (CYP) 3A4 and potent inducers of P-glycoprotein. This includes subjects who are on amiodarone or other contraindicated drugs. Refer to www.hep_druginteractions.org, the investigator manual and the investigator's brochure for detailed information.
8. Participation in other clinical trials within 3 months.
9. Any clinically significant findings or unstable condition during the screening, medical history or physical examination that, in the investigator's opinion, would compromise participation in this study. This could include patients with poorly controlled hypertension, asthma, diabetes, or other life-threatening conditions.
10. Current or history of use within the preceding 6 months of immunosuppressive or immune-modulating agents. Corticosteroid used to treat any medical condition are allowed if systemic for not more than 2 weeks or if topical.
11. History of solid organ or bone marrow transplantation.
12. Any prior DAA use or NS5A inhibitors therapy.
13. Patients with significant cardiovascular conditions including myocardial infarction within the previous 6 months or heart failure NYHA class III or IV; history of Torsade de pointes
14. HIV/HCV co-infected patients who are yet to receive stable antiretroviral therapy or for whom ART treatment initiation maybe scheduled during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
SVR12 | 12 weeks upon completion of treatment
  Sustained Virological Response (SVR) at week-12 post treatment, as evidenced by Hepatitis C Viral (HCV) ribonucleic acid (RNA) level less than the lower limit of quantification of 15 IU/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Radzi Abu Hassan, FRCP, Principal Investigator — Hospital Sultanah Bahiyah, Ministry of Health Malaysia
Locations (1):
- Hospital Sultanah Bahiyah, Alor Star, Kedah, Malaysia

IPD SHARING:
Plan to Share IPD: No